CLINICAL TRIAL: NCT01081509
Title: Survey and Follow-up of the Treatment Adherence and Medication Habits of Early Breast Cancer Patients on Adjuvant Hormonal Therapy With the Aromatase Inhibitor Arimidex
Brief Title: Survey Conducted Among Early Breast Cancer Patients Treated With Arimidex for Evaluation of Treatment Adherence
Acronym: ARIADNE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OHU-ARI-2010/1
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Breast Cancer
Keywords: adherence; early breast cancer; Arimidex; Therapy adherence
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to assess the patient's perception about and willingness to take his or her medication and the influencing factors interfering with taking medication.

ELIGIBILITY:
Inclusion Criteria:

* Early breast cancer
* Post menopausal
* Adjuvant hormonal Arimidex therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Early breast cancer patients on adjuvant aromatase inhibitor
Sampling Method: Probability Sample
Enrollment: 1077 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Percent of patients remaining adherent to therapy with Arimidex | Every 3 months

SECONDARY OUTCOMES:
Questionnaire for factors influencing adherence | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Zsolt Horvath, M.D., Ph.D., Principal Investigator — Hungarian National Institute of Oncology
Locations (25):
- Hungary (25):
  - Research Site, Balatonföldvár
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Dombóvár
  - Research Site, Gyöngyös
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Mosdós
  - Research Site, Nagyatád
  - Research Site, Nyíregyháza
  - Research Site, Orfű
  - Research Site, Pápa
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Szekszárd
  - Research Site, Szentes
  - Research Site, Székesfehérvár
  - Research Site, Szombathely
  - Research Site, Veszprém
  - Research Site, Zalaegerszeg
  - Research Site, Zirc